CLINICAL TRIAL: NCT04805515
Title: Impact of Nicotine Messaging on Nicotine Beliefs and Tobacco Use Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Andrea Villanti, Principal Investigator, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 00001374; R01DA051001 (NIH)
Record Dates: First submitted 2021-02-11; First posted 2021-03-18 (Actual); Results first posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Nicotine Dependence, Cigarettes
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Intervention Model Description: The intervention consists of 8 brief nicotine corrective public education messages delivered online. The messages will communicate misperceptions about nicotine's role in health harms as well as misperceptions that reduced nicotine content cigarettes are less harmful than tobacco cigarettes and that e-cigarettes contain less nicotine than tobacco cigarettes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nicotine Corrective Messages (Experimental): Participants in the nicotine corrective messages condition will receive 8 brief nicotine corrective public education messages delivered online during 4 waves of the 12 week study. The messages will communicate misperceptions about nicotine's role in health harms as well as misperceptions that reduced nicotine content cigarettes are less harmful than tobacco cigarettes and that e-cigarettes contain less nicotine than tobacco cigarettes.
  Interventions: Behavioral: Nicotine Corrective Messages
- Delayed Message Control (No Intervention): Participants in the control condition will be exposed to the nicotine corrective messages after the completion of the final assessment at the end of the 12 week study.

INTERVENTIONS:
Behavioral: Nicotine Corrective Messages — Messages communicating misperceptions of nicotine's role in health harms as well as misperceptions about reduced nicotine content cigarettes and e-cigarettes.
  Arms: Nicotine Corrective Messages

SUMMARY:
This is a 2-arm, randomized controlled, population based trial to test the impact of multiple exposures to brief nicotine corrective messages among adult tobacco cigarette smokers and non-smokers followed in waves over 12 weeks. The primary outcome, assessed at wave 1 (baseline), wave 2 (weeks 5-6), and wave 4 (weeks 11-13) is nicotine beliefs. Secondary outcomes assessed at the same time points include intention to use nicotine/tobacco products and nicotine/tobacco use.

DETAILED DESCRIPTION:
This is a 2-arm, randomized controlled, population based trial to test the impact of multiple exposures to brief nicotine corrective messages among adult tobacco cigarette smokers and non-smokers followed for 12 weeks. The primary outcome, assessed at wave 1 (baseline), wave 2 (weeks 5-6), and wave 4 (weeks 11-13) is nicotine beliefs. Secondary outcomes assessed at the same time points include intention to use nicotine/tobacco products and nicotine/tobacco use. All participants will be recruited from a US national consumer research panel. Eligible participants will be U.S. adults ages 18+ who are enrolled members of the partnering consumer research panel. The sample will include non-smokers and smokers, oversampling current smokers (defined as smoking 100+ lifetime cigarettes and now smoking all or some days) to ensure the proportion of smokers in the sample reflects the ~15 % population smoking prevalence among adults. Panel members will be contacted by email with a brief study description and link to an eligibility screener and online informed consent form. Eligible and interested participants will complete the baseline (Wave 1) survey measures of nicotine beliefs and intentions/use of nicotine and tobacco products, after which they will be randomly assigned in equal numbers to the nicotine corrective message (NCM) intervention condition or the delayed message control condition. After completing the baseline survey, participants in the NCM condition will receive their first exposure to the corrective messages. In the Wave 2 survey, all participants will complete measures of nicotine beliefs and intentions/use of nicotine and tobacco products. Participants in the NCM condition will then receive their second exposure to study messages. Only participants in the NCM condition will receive the Wave 3 survey, which involves the third exposure to study messages. The Wave 4 survey will include the fourth exposure to study messages for those in the NCM condition and the final assessment of nicotine beliefs and intentions/use of nicotine and tobacco products for all participants. Upon completion of the final assessment, participants in the control condition will be exposed to the nicotine corrective messages and all participants will be directed to resources on quitting smoking.

ELIGIBILITY:
Inclusion Criteria:

* US resident age 18+
* Member of the partnering consumer research panel conducting the survey
* Non-smokers and tobacco cigarette smokers

Exclusion Criteria:

* Age less than 18
* Not a member of the partnering consumer research panel conducting the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 794 (Actual)
Dates: Start 2021-02-12 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea C Villanti, PhD, MPH, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data from study surveys will be made available upon request and according to access criteria after completion of the study and publication of primary findings.
Time Frame: After completion of the study and publication of the primary findings, for a period up to 2 years.
Access Criteria: A data sharing agreement will be required for release of any data. Individuals requesting a copy of study data will need to submit a detailed research plan that includes the purpose of the proposed research, the variables required, the duration of the analysis phase, IRB approval with FWA information, investigator training in human subjects and other approvals specific to the individual datasets. They will also be required to submit a Data Protection Plan or Institutional Privacy Policy, describing the computing environment in which data will be managed and analyzed and how physical access to computing equipment will be controlled. Data will only be released once all IRB approvals and Human Subjects concerns have been addressed. The PI (A. Villanti) will be required to participate as an investigator on any project requiring data sharing.

REFERENCES:
- [Derived] Villanti AC, Peasley-Miklus C, Mercincavage M, Mays D, Donny EC, Cappella JN, Strasser AA. Effect of nicotine corrective messaging on nicotine-related beliefs in US adults: a randomised controlled trial. Tob Control. 2025 Apr 1;34(2):162-168. doi: 10.1136/tc-2023-058252. PMID 37989586

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were 794 U.S. English-speaking adults aged 18 and older recruited in spring 2021 from the AmeriSpeak® national consumer market research panel.
Period: Overall Study
Arm/Group | Nicotine Corrective Messages | Delayed Message Control
Started | 393 | 401
Wave 2 Survey | 313 | 318
Completed | 290 | 319
Not Completed | 103 | 82

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nicotine Corrective Messages | Delayed Message Control | Total
Number analyzed (Participants) | 393 | 401 | 794
Age, Customized [Count of Participants; unit: Participants]
  18-24 | 25 | 30 | 55
  25-34 | 78 | 84 | 162
  35-44 | 57 | 67 | 124
  45-54 | 61 | 62 | 123
  55-64 | 74 | 71 | 145
  65-74 | 68 | 67 | 135
  75+ | 30 | 20 | 50
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 186 | 214 | 400
  Male | 207 | 187 | 394
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 73 | 79 | 152
  White, non-Hispanic | 243 | 253 | 496
  Black, non-Hispanic | 40 | 37 | 77
  Asian, non-Hispanic | 13 | 6 | 19
  More than 1 race, non-Hispanic | 18 | 16 | 34
  Other race, non-Hispanic | 6 | 10 | 16
Any past 30-day tobacco use [Count of Participants; unit: Participants] | 80 | 89 | 169

OUTCOME MEASURES:

1. Primary Outcome: Nicotine Beliefs
Description: 3 items assessing nicotine false beliefs (range 3-11), 6 items assessing nicotine replacement therapy (NRT) false beliefs (range 4-20), 4 items assessing e-cigarette false beliefs (range 2-14), 11 items assessing reduced nicotine content (RNC) cigarette false beliefs (range 14-45), and two items assessing beliefs about additive-free and organic tobacco products. Higher scale scores indicate a higher number of false beliefs.
Time Frame: Wave 4 (weeks 11-13)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nicotine Corrective Messages | Delayed Message Control
Number analyzed (Participants) | 290 | 319
score on a scale
  Nicotine false beliefs (range 3-11) | 7.5 (2.3) | 7.8 (2.1)
  NRT false beliefs (range 4-20) | 10.9 (2.8) | 11.3 (2.8)
  E-cigarette false beliefs (range 2-14) | 8.9 (2.2) | 9.2 (2.1)
  Reduced nicotine content cigarette false beliefs (range 14-45) | 29.8 (4.7) | 30.3 (4.1)

2. Secondary Outcome: Intention to Use Nicotine/Tobacco Products
Description: Four items assessing intention to use tobacco cigarettes, e-cigarettes, NRT, and RNC cigarettes during the next 12 months. Adapted from PhenX Toolkit- Susceptibility to Tobacco Products, response options Definitely Yes; Probably Yes; Probably Not; Definitely Not. Outcomes reported for participants reporting Definitely Yes or Probably Yes to each item.
Time Frame: Wave 4 (weeks 11-13)
Population: The number of participants analyzed differs from the overall number due to item non-response.
Measure: Count of Participants; unit: Participants
Arm/Group | Nicotine Corrective Messages | Delayed Message Control
Number analyzed (Participants) | 290 | 319
Participants
  Cigarette: number analyzed (Participants) | 289 | 319
  Cigarette | 56 | 50
  E-cigarette/vape: number analyzed (Participants) | 290 | 317
  E-cigarette/vape | 20 | 27
  Nicotine replacement product: number analyzed (Participants) | 290 | 318
  Nicotine replacement product | 20 | 23
  Low nicotine cigarette | 28 | 15

3. Secondary Outcome: Tobacco Use
Description: Number of days used tobacco in the past 30 days. Days used summed across eight different nicotine/tobacco products (e.g., tobacco cigarettes, e-cigarettes, cigars, NRT, RNC cigarettes).
Time Frame: Wave 4 (weeks 11-13)
Population: Analyses restricted to participants who reported any past 30-day tobacco use at baseline.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Nicotine Corrective Messages | Delayed Message Control
Number analyzed (Participants) | 80 | 89
Days | 18.6 (16.5) | 18.4 (18.7)

4. Other Pre Specified Outcome: Attitudes About Nicotine
Description: Three items on nicotine-related attitudes using semantic differentials across five-point Likert scales. 'Using Nicotine is:' Safe (1) - Dangerous (5); Positive (1) - Negative (5); Good (1) - Bad (5).
Time Frame: Wave 4 (weeks 11-13)
Population: The analytic sample differs from the overall sample due to item non-response.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nicotine Corrective Messages | Delayed Message Control
Number analyzed (Participants) | 290 | 319
score on a scale
  Safe to Dangerous: number analyzed (Participants) | 290 | 317
  Safe to Dangerous | 4.4 (0.9) | 4.5 (0.8)
  Positive to Negative: number analyzed (Participants) | 288 | 317
  Positive to Negative | 4.6 (0.7) | 4.5 (0.8)
  Good to Bad: number analyzed (Participants) | 289 | 317
  Good to Bad | 4.6 (0.8) | 4.6 (0.8)

5. Other Pre Specified Outcome: Nicotine Related Norms
Description: Two items: "How would you describe most people's opinion of using nicotine?" and "Thinking about the people who are important to you, how would you describe their opinion on using nicotine?" with five-point Likert scale responses ranging from "very negative" (1) to "very positive" (5). Higher scores indicate positive norms of using nicotine.
Time Frame: Wave 4 (weeks 11-13)
Population: The analytic sample differs from the overall sample due to item non-response.
Measure: Mean (Standard Deviation); unit: score on a Likert scale
Arm/Group | Nicotine Corrective Messages | Delayed Message Control
Number analyzed (Participants) | 290 | 319
score on a Likert scale
  People who are important to you: number analyzed (Participants) | 289 | 319
  People who are important to you | 1.9 (0.9) | 2.1 (1.0)
  Most people: number analyzed (Participants) | 290 | 318
  Most people | 2.1 (0.7) | 2.2 (0.8)

6. Other Pre Specified Outcome: Behavioral Control
Description: One item assessing confidence to resist smoking cigarettes when others are smoking (1=not at all confident to 4=very confident).
Time Frame: Wave 4 (weeks 11-13)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nicotine Corrective Messages | Delayed Message Control
Number analyzed (Participants) | 290 | 318
score on a scale | 3.6 (0.8) | 3.6 (0.9)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Nicotine Corrective Messages | Delayed Message Control
All-Cause Mortality (participants affected / at risk) | 0/393 | 0/401
Serious Adverse Events (participants affected / at risk) | 0/393 | 0/401
Other Adverse Events (participants affected / at risk) | 0/393 | 0/401

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-18): https://cdn.clinicaltrials.gov/large-docs/15/NCT04805515/Prot_SAP_000.pdf